CLINICAL TRIAL: NCT04231435
Title: A Phase 1, Open-label Study to Evaluate the Influence of Fedratinib on the Pharmacokinetics of Transporter Probe Substrates (Digoxin, Rosuvastatin, and Metformin) in Healthy Adult Subjects
Brief Title: Influence of Fedratinib on the Pharmacokinetics of the Transporter Probe Substrates Digoxin, Rosuvastatin, and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-CP-003; U1111-1245-6233 (Other: WHO)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Adult Subjects; Fedratinib; Drug Interactions; Transporters
MeSH Terms: interventions — fedratinib; Digoxin; Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Administration (Experimental): All subjects will receive the following oral doses of IP following an overnight fast in the fixed-sequence below:
  * Day 1 (Period 1): 1 × 0.25-mg digoxin tablet, 1 × 10-mg rosuvastatin tablet, and 1 × 1000-mg metformin tablet.
  * Day 7 (Period 2): 6 × 100-mg fedratinib capsules PLUS (after approximately 1 hour from the time of fedratinib administration) 1 × 0.25 mg digoxin tablet, 1 × 10-mg rosuvastatin tablet, and 1 × 1000-mg metformin tablet.
  Interventions: Drug: Fedratinib; Drug: Digoxin; Drug: Rosuvastatin; Drug: Metformin

INTERVENTIONS:
Drug: Fedratinib — Oral
Drug: Digoxin — Oral
Drug: Rosuvastatin — Oral
Drug: Metformin — Oral

SUMMARY:
This is a nonrandomized, fixed-sequence, open-label study to evaluate the effect of a single dose of fedratinib on the PK, safety, and tolerability of single doses of digoxin, rosuvastatin, and metformin in healthy subjects. The subjects will participate as follows:

* Screening phase
* Treatment phase (includes baseline)
* Follow-up telephone call Subjects will be screened for eligibility during the screening phase. Subjects who meet all inclusion criteria and none of the exclusion criteria will return to the clinical site on Day -1 for protocol-specified assessments, and will be domiciled at the clinical site from Day -1 through the morning of Day 22.

During the study, blood samples will be collected at prespecified times for PK and PD. Urine samples will be collected at prespecified times for urinary PK evaluation of metformin. Subject safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject must be willing and able to communicate with the Investigator and adhere to the study visit schedule and other protocol requirements.
3. Subject is male or female of any race ≥ 18 to ≤ 65 years of age at the time of signing the ICF.
4. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level in the post-menopausal range according to the laboratory used at Screening).
5. Females of childbearing potential (FCBP1) must:

   1. Have a negative pregnancy test as verified by the investigator at Screening and Baseline (prior to starting study treatment). She must agree to ongoing pregnancy testing during the course of the study, as applicable, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use, and be able to comply with, any one of the following highly effective contraception methods without interruption, beginning at least 14 days prior to starting investigational product (IP), during the study treatment, and for at least 30 days after the last dose of IP. - Intrauterine device (IUD; non-hormonal only); tubal ligation; or a partner with a vasectomy. The chosen form of birth control must be effective by the time the subject receives the first dose of IP.
6. Male subjects must:

   a. Practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made from natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while receiving study treatment, and for at least 30 days after the last dose of IP, even if he has undergone a successful vasectomy.
7. Must have a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
8. Must be healthy, as determined by the Investigator on the basis of medical history, physical examination (PE), clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG) at screening and check-in (Day -1), as applicable:

   Aspartate aminotransferase (AST), ALT, and total bilirubin must be at or below the upper limit of the reference range on or before check-in (Day -1). Other clinical laboratory results must be either within normal range or deemed not clinically significant by the Investigator. Any out of range lab tests may be repeated up to 1 time during Screening and up to 1 time at check-in per Investigator discretion to confirm eligibility.
9. Must be afebrile (febrile is defined as ≥ 38°C or 100.3°F).
10. Supine systolic blood pressure (BP) must be in the range of 90 to 140 mmHg (inclusive), supine diastolic BP must be in the range of 50 to 90 mmHg (inclusive), and pulse rate must be in the range of 45 to 100 bpm (inclusive) at screening.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening; male subjects must have a corrected QT interval using Fridericia's formula (QTcF) value ≤ 430 msec and females must have a QTcF value ≤ 450 msec. An ECG may be repeated up to 2 times, and the average of the QTcF values will be used to determine subject eligibility.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History (within 3 years prior to Screening) of any clinically significant neurological, GI, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders as determined by the Investigator.
2. Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable).
3. Subject has prior history of Wernicke's Encephalopathy (WE).
4. Subject has signs or symptoms of WE (eg, ataxia, ocular paralysis, or cerebellar signs) without documented exclusion of WE by thiamine level and brain magnetic resonance imaging (MRI).
5. Subject has thiamine deficiency, defined as thiamine levels in whole blood below normal range according to institutional standard.
6. Subject has an estimated glomerular filtration rate (GFR) of <90 mL/min/1.73 m2 based on the 4-variable Modification of Diet in Renal Disease (MDRD) equation.
7. Use of any prescribed systemic or topical medication, including vaccines, within 30 days of the first dose administration (with the exception of any palonosetron administered for purposes of this study).
8. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 14 days of the first dose administration (with the exception of acetaminophen up to 2 grams/day for no more than 3 consecutive days to treat minor illness or headache [per Investigator judgment]).
9. Use of any metabolic enzyme or relevant transporter inhibitors or inducers that would affect the relevant drugs within 30 days of the first dose administration unless determined by the Investigator that there will be no impact on the study integrity or subject safety.

   The Indiana University "P450 Drug Interaction Table" should be used to determine inhibitors and/or inducers of metabolic enzymes (http://medicine.iupui.edu/clinpharm/ddis/table/aspx). The Sponsor should be contacted for questions about potential drug-drug interactions and exclusions/prohibitions when necessary.
10. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
11. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion (eg, bariatric procedure, cholecystectomy).

    Appendectomy is acceptable.
12. Donated blood or plasma within 8 weeks before the first dose administration.
13. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing or positive drug screening test reflecting consumption of illicit drugs.
14. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing or positive alcohol screen.
15. Known to have serum hepatitis; known to be a carrier of the hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), or hepatitis C antibody (HCV Ab); have a positive result to the test for hepatitis B or hepatitis C virus at screening or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening. Subjects whose results are compatible with prior immunization (including natural and vaccination) against hepatitis B may be included at the discretion of the Investigator.
16. Subject smokes > 10 cigarettes per day, or equivalent in other tobacco products, more frequently than 8 weeks prior to Screening (self-reported).
17. History of multiple drug allergies (ie, 2 or more).
18. Allergic to or hypersensitive to any of the drugs used in the study.
19. Has any medical condition, medical history, or use of concomitant medication that is contraindicated in the applicable drug labeling.

    Note: Subjects having a history of intolerability or hypersensitivity to selective serotonin reuptake inhibitors, monoamine oxidase-B inhibitors, or serotonin-norepinephrine reuptake inhibitors that are suggestive of serotonin syndrome or related AE are not eligible for study participation.
20. Female subject who is pregnant or breastfeeding.
21. Subject is part of the clinical staff personnel or a family member of the clinical site staff.
22. Subject has a hypersensitivity to palonosetron.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax (Digoxin, Rosuvastatin and Metformin | 96 hours
  Maximum observed plasma concentration
Pharmacokinetic - AUC (Digoxin, Rosuvastatin and Metformin | 96 hours
  Area under the curve
Pharmacokinetic - CLr | 48 hours
  Renal Clearance
Analysis of Glucose AUC after OGTT using linear trapezoidal method | 3 hours
  Area under the curve

SECONDARY OUTCOMES:
Adverse Events (AEs) | From the time the ICF is signed until study completion and up to 30 days after the last dose of IP
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopolous, M.D., Study Director — Celgene
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Ogasawara K, Wood-Horrall RN, Thomas M, Thomas M, Liu L, Liu M, Xue Y, Surapaneni S, Carayannopoulos LN, Zhou S, Palmisano M, Krishna G. Impact of fedratinib on the pharmacokinetics of transporter probe substrates using a cocktail approach. Cancer Chemother Pharmacol. 2021 Dec;88(6):941-952. doi: 10.1007/s00280-021-04346-7. Epub 2021 Sep 3. PMID 34477937